CLINICAL TRIAL: NCT07130227
Title: The Effect of MBRS-Based Psychoeducation on Anger Management and Functional Recovery in Patients With Schizophrenia
Brief Title: MBRS-Based Psychoeducation in Patients With Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Mine CENGİZ, Lecturer Physician, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: MCENGİZ5
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Mindfulness Training
Keywords: mindfulness; Schizophrenia; Psychoeducation; Nursing
MeSH Terms: conditions — Schizophrenia | interventions — mycophenolic adenine dinucleotide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (24):
- Session 1: Preparatory Session (Experimental): *Meeting the patients *Introducing the content of mindfulness-based stress reduction training *Emphasizing the importance of regular and timely attendance at training *Determining training dates *Sharing individuals' experiences and expectations
  Interventions: Other: Session 1: Preparatory Session
- Session 2: Mindfulness (Experimental): *What is mindfulness? *Being aware of daily activities. *Raisin meditation.
  Interventions: Other: Session 2: Mindfulness
- Session 3: Our Perspectives on Ourselves and the World (Experimental): *Breathing meditation. *Habit Breaker: Watching the Sky.
  Interventions: Other: Session 3: Our Perspectives on Ourselves and the World
- Session 4: Body Scan *Body scan meditation. (Experimental): *Ten-finger gratitude practice. *Habit Breaker: Spending some time in nature.
  Interventions: Other: Session 4: Body Scan *Body scan meditation.
- Session 5: Recognizing Schizophrenia (Experimental): *What is schizophrenia? *What are its symptoms? *What does treatment involve?
  Interventions: Other: Session 5: Recognizing Schizophrenia
- Session 6: Mindful Movement (Experimental): *Mindfulness movement meditation practice *
  Interventions: Other: Session 6: Mindful Movement
- Session 7: Mindful Breathing (Experimental): *Breathing meditation
  Interventions: Other: Session 7: Mindful Breathing
- Session 8: Treatment Evaluation (Experimental): *The importance of medication *Things to consider when using medication *Side effects of medication *What is a flare-up in schizophrenia? *What are the precursor symptoms?
  Interventions: Other: Session 8: Treatment Evaluation
- Session 9: Mindful Thinking (Experimental): *Sounds and thoughts meditation *Cinema activity.
  Interventions: Other: Session 9: Mindful Thinking
- Session 10: Coping with Anger (Experimental): *What is anger? *What are its symptoms? *What are the coping methods?
  Interventions: Other: Session 10: Coping with Anger
- Session 11: Coping with Difficult Emotions (Experimental): *Facing Difficulties meditation
  Interventions: Other: Session 11: Coping with Difficult Emotions
- Session 12: Mindful Communication (Experimental): *Communication & mindful communication *The importance of communication skills *Fundamentals of communication, self-language practice *Ways to prevent communication accidents
  Interventions: Other: Session 12: Mindful Communication
- Session 13: Different Connections (Experimental): *Breathing meditation. *Habit Breaker: Thought and Emotional Play.
  Interventions: Other: Session 13: Different Connections
- Session 14: The Joy of the Small Things (Experimental): *Treasure Treasure Meditation *Habit Breaker: Letter to Self.
  Interventions: Other: Session 14: The Joy of Small Things
- Session 15: Dwelling on the Past or Living in the Present? (Experimental): *Friendship-Building Meditation *Habit Breaker: Random Acts of Kindness.
  Interventions: Other: Session 15: Dwelling on the Past or Living in the Present?
- Session 16: Evaluation *Reinforcing What Has Been Learned. (Experimental): *Evaluating the Program. *Obtaining Feedback.
  Interventions: Other: Session 16: Evaluation
- Group 2: 2: Recognizing the Illness (Active Comparator): *What is schizophrenia? *What are its symptoms? *What does treatment involve?
  Interventions: Other: Session 2: Group 2, Recognizing the Illness
- Group 2: Session 3: Evaluating Treatment (Active Comparator): *Considerations regarding medication use *Side effects of medication use *Exacerbations in schizophrenia *Premonitory symptoms.
  Interventions: Other: Session 3: Group 2, Treatment Evaluation
- Group 2: Session 4: *What is anger? (Active Comparator): *What are the symptoms of anger? *What are the methods for coping with anger?
  Interventions: Other: Session 4: Group 2, What is anger?
- Group 2: Session 5: Communication *What is communication? (Active Comparator): *The importance of communication. *Fundamentals of communication, self-language practice *Ways to prevent communication difficulties.
  Interventions: Other: Session 5: Group 2, Communication
- Group 2: Session 6: What is relaxation? (Active Comparator): What is progressive relaxation. Relaxation CD introduction
  Interventions: Other: Session 6: Group 2, What is relaxation?
- Group 2: Session 7: Relaxation (Active Comparator): Performing the relaxation CD with patients
  Interventions: Other: Session 7: Group 2, Relaxation
- Group 2: Session 8: Evaluation (Active Comparator): *Reinforcement of what has been learned. *Evaluation of the program. *Receiving feedback
  Interventions: Other: Session 8: Group 2, Evaluation
- Group 2: Session 1: Preparatory Session (Active Comparator): *Meeting the patients *Introducing the content of psychoeducation *Emphasizing the importance of regular and timely attendance at training *Determining training dates *Sharing individuals' experiences and expectations
  Interventions: Other: Session 1: Group 2, Preparation Session

INTERVENTIONS:
Other: Session 1: Preparatory Session — *Meeting the patients *Introducing the content of mindfulness-based stress reduction training *Emphasizing the importance of regular and timely attendance at training *Determining training dates *Sharing individuals' experiences and expectations
  Arms: Session 1: Preparatory Session
Other: Session 2: Mindfulness — *What is mindfulness? *Being aware of daily activities. *Raisin meditation.
  Arms: Session 2: Mindfulness
Other: Session 3: Our Perspectives on Ourselves and the World — *Breathing meditation. *Habit Breaker: Watching the Sky.
  Arms: Session 3: Our Perspectives on Ourselves and the World
Other: Session 4: Body Scan *Body scan meditation. — *Ten-finger gratitude practice. *Habit Breaker: Spending some time in nature.
  Arms: Session 4: Body Scan *Body scan meditation.
Other: Session 5: Recognizing Schizophrenia — *What is schizophrenia? *What are its symptoms? *What does treatment involve?
  Arms: Session 5: Recognizing Schizophrenia
Other: Session 6: Mindful Movement — *Mindfulness movement meditation practice *
  Arms: Session 6: Mindful Movement
Other: Session 7: Mindful Breathing — *Breathing meditation *
  Arms: Session 7: Mindful Breathing
Other: Session 8: Treatment Evaluation — *The importance of medication *Things to consider when using medication *Side effects of medication *What is a flare-up in schizophrenia? *What are the precursor symptoms?
  Arms: Session 8: Treatment Evaluation
Other: Session 9: Mindful Thinking — *Sounds and thoughts meditation *Cinema activity.
  Arms: Session 9: Mindful Thinking
Other: Session 10: Coping with Anger — *What is anger? *What are its symptoms? *What are the coping methods?
  Arms: Session 10: Coping with Anger
Other: Session 11: Coping with Difficult Emotions — *Facing Difficulties meditation *
  Arms: Session 11: Coping with Difficult Emotions
Other: Session 12: Mindful Communication — *Communication & mindful communication *The importance of communication skills *Fundamentals of communication, self-language practice *Ways to prevent communication accidents
  Arms: Session 12: Mindful Communication
Other: Session 13: Different Connections — *Breathing meditation. *Habit Breaker: Thought and Emotional Play.
  Arms: Session 13: Different Connections
Other: Session 14: The Joy of Small Things — *Treasure of Pleasure Meditation *Habit Breaker: Letter to Self.
  Arms: Session 14: The Joy of the Small Things
Other: Session 15: Dwelling on the Past or Living in the Present? — *Friendship-Building Meditation *Habit Breaker: Random Acts of Kindness.
  Arms: Session 15: Dwelling on the Past or Living in the Present?
Other: Session 16: Evaluation — *Reinforcing What Has Been Learned. *Evaluating the Program. *Obtaining Feedback.
  Arms: Session 16: Evaluation *Reinforcing What Has Been Learned.
Other: Session 1: Group 2, Preparation Session — *Meeting Patients *Introducing the Content of Psychoeducation *Emphasizing the Importance of Regular and Timely Attendance at Training *Determining Training Dates *Sharing Individuals' Experiences and Expectations
  Other Names: Active Participant
  Arms: Group 2: Session 1: Preparatory Session
Other: Session 2: Group 2, Recognizing the Illness — *What is Schizophrenia? *What are its Symptoms? *What Does Treatment Include?
  Arms: Group 2: 2: Recognizing the Illness
Other: Session 3: Group 2, Treatment Evaluation — *Things to Consider When Using Medication *Side Effects of Medication *Exacerbation of Schizophrenia *Precursor Symptoms.
  Arms: Group 2: Session 3: Evaluating Treatment
Other: Session 4: Group 2, What is anger? — *What are the symptoms of anger? *What are the methods for coping with anger?
  Arms: Group 2: Session 4: *What is anger?
Other: Session 5: Group 2, Communication — *What is communication? *The importance of communication. *Fundamentals of communication, working on "I" language. *Ways to prevent communication difficulties.
  Arms: Group 2: Session 5: Communication *What is communication?
Other: Session 6: Group 2, What is relaxation? — What is progressive relaxation? Introducing a relaxation CD
  Arms: Group 2: Session 6: What is relaxation?
Other: Session 7: Group 2, Relaxation — Practicing the relaxation CD with patients
  Arms: Group 2: Session 7: Relaxation
Other: Session 8: Group 2, Evaluation — *Reinforcing what has been learned. *Evaluating the program. *Obtaining feedback
  Arms: Group 2: Session 8: Evaluation

SUMMARY:
This study aimed to determine the effects of mindfulness-based stress reduction training on anger management and functional recovery in patients with schizophrenia. The study will be conducted at a CMHC in Ağrı province between May and August 2021. At the CMHC, community-based mental health services are provided to patients with severe mental disorders (schizophrenia, bipolar disorder) who are in remission as assessed by a psychiatrist. The study is planned to be conducted with patients who meet the study criteria, without using a sample selection method. Patients over the age of 18 registered with CMHC and followed with a diagnosis of schizophrenia were contacted by phone and invited to CMHC. The study was conducted with patients who met the inclusion criteria and agreed to participate (psychoeducational group, mindfulness group, control group). Data will be collected using the Descriptive Characteristics Form, the State and Trait Anger Inventory, and the SILO. The mindfulness group received 16 sessions of MBRS training, and the psychoeducational group received an 8-session psychoeducational program. The control group received no intervention. The study sample size was calculated using the GPower computer program. Power analysis at α=0.05 yielded an effect size of 150, 153 (d=0.8), and the study had 90% power. Therefore, it was calculated that a minimum of 68 patients should be included in the sample.

DETAILED DESCRIPTION:
Study data were collected by the researcher through face-to-face interviews. The study included individuals diagnosed with schizophrenia who met the inclusion criteria (registration in a CMHC, having a diagnosis of schizophrenia, willingness to participate in the study, and openness to communication and collaboration). Pre-test measurement instruments were administered to the participants. The mindfulness group then received 16 sessions of MBRS training, and the psychoeducation group received an 8-session psychoeducation program. The control group received no intervention. Post-test data were collected following the training sessions.

ELIGIBILITY:
Inclusion Criteria:

* Being registered with a CMHC
* Being diagnosed with schizophrenia
* Being between the ages of 18 and 60
* Being willing to participate in the study
* Being open to communication and cooperation
* Being in remission

Exclusion Criteria:

* Not being open to communication and cooperation

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2021-03-30 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Personal Information Form | up to 1 day
  This form consists of a total of eight questions (age, gender, marital status, education level, duration of illness, income, family history of mental illness, and employment status) developed by the researcher based on literature and includes the sociodemographic characteristics of the patients

SECONDARY OUTCOMES:
The State-Trait Anger Scale (STAS) | up to 1 day
  This is a self-report scale measuring the feeling and expression of anger. It was developed by Spielberger et al., and its Turkish validity and reliability study was conducted by Özer. The Cronbach's alpha obtained in this study was 0.84. The scale is a four-point Likert-type scale consisting of four subscales: anger-in, anger-out, anger control, and trait anger, and 34 items. High scores on the trait anger dimension indicate high anger levels, high scores on the anger control dimension indicate that anger can be controlled, high scores on the anger-out dimension indicate that anger is easily expressed, and high scores on the anger-in dimension indicate that anger is suppressed.

OTHER OUTCOMES:
Functional Recovery Scale in Schizophrenia (FRS) | up to 1 day
  The Functional Recovery Scale in Schizophrenia (FRS) was developed by Llorca et al. in 2009. The scale's validity and reliability in Turkey were conducted by Emiroğlu in 2009. The validity and reliability coefficient of the scale was determined to be 0.94. In this study, the Chronbach's alpha coefficient was determined to be 0.91. It is a 5-point Likert-type scale consisting of 19 items and 4 subscales. As the scores on the scale increase, the level of functional recovery increases. Dimensions: Social Functioning (7 items), Health and Treatment (4 items), Daily Living Skills (6 items), Occupational Functioning (2 items). The lowest score that can be obtained from the scale is 19, the highest score is 95.

CONTACTS AND LOCATIONS:
Overall Officials: Mine Cengiz lecturer doctor, Principal Investigator — Ataturk University
Locations (1):
- Ataturk University Faculty of Nursing, Erzurum, Yakutiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided